CLINICAL TRIAL: NCT01342055
Title: Phase I Study of Apetrol ES and Megace® in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety Study of Apetrol ES in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-ESCL002
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 : Megace 800mg - Apetrol ES 650mg - Apetrol ES 675mg (Experimental)
  Interventions: Drug: Apetrol ES
- Group 2 : Apetrol ES 650mg - Apetrol ES 675mg -Megace 800mg (Experimental)
  Interventions: Drug: Apetrol ES
- Group 4: Megace 800mg - Apetrol ES 675mg - Apetrol ES 650mg (Experimental)
  Interventions: Drug: Apetrol ES
- Group 5: Apetrol ES 650mg - Megace 800mg - Apetrol ES 675mg (Experimental)
  Interventions: Drug: Apetrol ES
- Group 3: Apetrol ES 675mg - Apetrol ES 650mg - Megace 800mg (Experimental)
  Interventions: Drug: Apetrol ES
- Group 6 : Apetrol ES 675mg - Megace 800mg - Apetrol ES 650mg (Experimental)
  Interventions: Drug: Apetrol ES

INTERVENTIONS:
Drug: Apetrol ES — sequences of administered drugs

SUMMARY:
A Randomized, Open Label, Single dose, Cross-over, Phase I Trial to Investigate Safety and Pharmacokinetics of Apetrol ES and Megace® under Fed Conditions in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Is a healty male between 20 and 55 years old
* Has BMI result between 19 and 26 kg/m2 at screening
* Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Agrees to use an adequate means of contraception during clinical trials

Exclusion Criteria:

* Has had a serious illness or medical condition(s) regarding liver, kidney, gastrointestines, pulmonary systems, etc.
* Has had a medical history of gastrointestinal diseases which might affect drug absorption (i.e. Crohn's disease, ulcer) or surgical history.
* Is allergic against Megestrol acetate or other drugs (Aspirin, NSAIDs, Antibiotics, etc.) or against foods, or has an clinically serious allergic history

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cmax, AUClast | Day 34

SECONDARY OUTCOMES:
AUCinf, Tmax, t1/2(beta) | Day 34

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim YH, Choi HY, Jin S, Noh YH, Kim MJ, Park HJ, Lim HS, Bang K, Lee SH, Bae KS. Tolerability and pharmacokinetics of two formulations of megestrol acetate under fed conditions in healthy volunteers. Clin Ther. 2015 Feb 1;37(2):439-47. doi: 10.1016/j.clinthera.2014.09.022. Epub 2014 Oct 23. PMID 25450470